CLINICAL TRIAL: NCT03982771
Title: Bortezomib, Cyclophosphamide and Dexamethasone (BCD) in Newly Diagnosed Idiopathic Multicentric Castleman's Disease (iMCD) : a Prospective, Single-center, Single-arm, Phase-II Pilot Trial
Brief Title: BCD Regimen in Newly Diagnosed Idiopathic Multicentric Castleman's Disease (iMCD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Jian Li, Professor in hematology, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZS-1892
Record Dates: First submitted 2019-05-03; First posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Idiopathic Multicentric Castleman's Disease
Keywords: Idiopathic Multicentric Castleman's Disease; BCD Regimen; Efficacy; Safety
MeSH Terms: conditions — Multi-centric Castleman's Disease | interventions — Bortezomib; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: This will be a single center, single arm, phase-II pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BCD regimen (Experimental): Bortezomib, cyclophosphamide and dexamethasone (the BCD regimen) would be utilized in newly diagnosed iMCD (idiopathic Multicentric Castleman's disease) patients
  Interventions: Drug: Bortezomib; Drug: Cyclophosphamide; Drug: Dexamethason

INTERVENTIONS:
Drug: Bortezomib — -Bortezomib: 1.3mg/m2 subcutaneous injection on Day 1,8,15,22 every month for 9 months; And maintained with 1.3mg/m2 subcutaneous injection every two weeks from Month 9 to 21;
Drug: Cyclophosphamide — -Cyclophosphamide: (oral) 300mg/m2 on Day 1, 8, 15, 22 every month for 9 months;
Drug: Dexamethason — Dexamethasone: (oral) 40mg on Day 1,8,15,22 every month for 9 months; and maintained with 20mg (oral) every two weeks from Month 9 to 21.

SUMMARY:
To explore the effectiveness and safety of bortezomib, cyclophosphamide and dexamethasone (BCD regimen) in newly diagnosed idiopathic Multicentric Castleman's disease (iMCD) patients.

DETAILED DESCRIPTION:
This will be a single center, open-labeled, single arm, phase-II pilot study. The treatment and the response evaluation phase will last from the time of enrollment up to 21 months (evaluation will be carried out every 3 months in the first 9 months and every 6 months from Month 9 to Month 21). The maintenance and follow-up phase to assess for progression of disease will last from 21 months to 45 months after enrollment (evaluation will be carried out every 12 months). The total study duration will be 4 years after the last patient starts study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Demography: ≥18 years, all race/ethnic groups in China;
2. Newly diagnosed and previously untreated (patients are allowed to have received oral prednisone for up to 1 week before enrollment) symptomatic iMCD patients (symptomatic disease is defined by the presence of clinical symptoms with the NCI-CTCAE grading ≥1 that are attributable to the disease, and for which treatment is indicated; iMCD diagnosis is based on the international consensus diagnostic criteria);
3. Clinical laboratory values meeting these criteria at screening: absolute neutrophil count ≥ 1·0 x 109/L, Platelets ≥ 50 x 109/L, Alanine aminotransferase (ALT) within 2·5 x upper limit of normal (ULN); total bilirubin within 2·5 x ULN; estimated glomerular filtration rate (according to MDRD formula) <15ml/min;
4. Women of childbearing potential must agree to use birth control measures during the study and for at least 3 months after receiving the last dose of study agent, and must have a negative pregnancy test at screening period. Men must agree to use birth control measures during the study and for at least 3 months after receiving the last dose of study agent;
5. Informed consent must be signed.

Exclusion Criteria:

1. age under 18 years;
2. Immunosuppressive or anti-neoplastic drugs within the last 3 months;
3. serious diseases including malignancy;
4. Plan to have babies within 1 year after enrollment (for women and men), or pregnancy / breast-feeding (for women);
5. Known hypersensitivity to study agents;
6. Active infection requiring systemic treatment;
7. Other severe concurrent disease (eg. uncontrolled diabetes, symptomatic coronary heart disease) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study;
8. Unwilling or unable to provide informed consent;
9. Unwilling to return for follow-up at PUMCH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall response | 12 months after the last patient begins study treatment.
  Overall response is composed by biochemical, lymph node and symptom response, is the primary outcome of this study. According to the CDCN response criteria, an overall CR (complete response) requires a complete biochemical, lymph node, and symptomatic response; and overall PR (partial response) requires nothing less than a PR across all categories, but not meeting criteria for CR; an overall SD (stable disease) requires no PD (progression disease) in any of the categories and not meeting the criteria for CR or PR; an overall PD occurs when any category has a PD.

SECONDARY OUTCOMES:
Time to initial response | 12 months after the last patient begins study treatment.
  defined as the time to achieve the first PR or CR. This outcome can be further divided into time to initial overall response, time to initial symptomatic response, time to initial biochemical response, time to initial lymph node response
Time to best response | 12 months after the last patient begins study treatment.
  defined as the time to achieve the best response (either PR or CR). This outcome can be further divided into time to best overall response, time to best symptomatic response, time to best biochemical response, time to best lymph node response;
Progression-free survival (PFS) | 12 months after the last patient begins study treatment.
  defined as the time to disease PD
Overall survival (OS) | 12 months after the last patient begins study treatment.
  defined as the time to patients' death
Change in PHQ-9 score | From Day 1 of the BCD treatment until 12 months after the treatment
  PHQ-9 score (Patient Health Questionnaire scale-9) is a nine-item self-administered instrument to assess depressive symptoms which incorporates the DSM-IV (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition) classification for major depressive disorder. Each item is scored 0 - 3, which results in a range of scores between 0 and 27. PHQ-9 scores are interpreted as follows: (1) score <5, no depression; (2) score 5 - 9, mild depression; (3) score 10 - 14, moderate depression; (4) score 15 - 19, moderately severe depression; and (5) score 20 - 27,severe depression.
Change in hemoglobin level | From baseline until 12 months after the treatment
  hemoglobin with g/L as unit of measure
Change in IL-6 (interleukin-6) | From baseline until 12 months after the treatment
  IL-6 level with pg/ml as unit of measure
Change in CRP | From baseline until 12 months after the treatment
  CRP (c-reactive protein) level with mg/L as unit of measure
Change in ESR | From baseline until 12 months after the treatment
  ESR (eerythrocyte sedimentation rate) level with mm/h as unit of measure
Change in IgG level | From baseline until 12 months after the treatment
  IgG (immunoglobin G) level with g/L as unit of measure
Change in MCD-related overall symptom score | From baseline until 12 months after the treatment
  Change of MCD symptom scores. MCD symptom score (MCD disease related overall symptom score) is a 34-item score based on NCI-CTCAE (V4.0) adverse events. Each item is scored 0-5, which results in a range of scores between 0 and 170. More scores indicate more severe disease activity.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 ( ≥1 grade) | 12 months after the last patient begins study treatment.
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 (patients with grades ≥1 would be included)
Number of participants with treatment-related serious adverse events as assessed by CTCAE v4.0 ( ≥3 grade) | 12 months after the last patient begins study treatment
  Number of participants with treatment-related serious adverse events as assessed by CTCAE v4.0 (patients with grades ≥3 would be included)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao H, Zhang MY, Shen KN, Feng J, Cao XX, Duan MH, Zhou DB, Zhang L, Li J. A phase 2 prospective study of bortezomib, cyclophosphamide, and dexamethasone in patients with newly diagnosed iMCD. Blood. 2023 May 25;141(21):2654-2657. doi: 10.1182/blood.2023020009. No abstract available. PMID 36928290